CLINICAL TRIAL: NCT06875180
Title: The Effect of Tele-Rehabilitation on Pain, Kinesiophobia and Disability in Patients With Chronic Non-Specific Low Back Pain
Brief Title: The Effects of Tele-Rehabilitation in Patients With Chronic Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pınar Kuyulu (Other)
Responsible Party: Sponsor-Investigator, Pınar Kuyulu, Pınar Kuyulu Haksal, PhD(c), Sanko University
Organization: Sanko University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/25
Record Dates: First submitted 2025-01-29; First posted 2025-03-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Non-Spesific Chronic Low Back Pain
Keywords: Chronic non-specific low back pain; telerehabilitation; McKenzie; disability; kinesiophobia; pain; range of motion
MeSH Terms: conditions — Kinesiophobia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation group (Experimental): Tele-rehabilitation exercise was applied to this group.
  Interventions: Other: Tele-rehabilitation exercise
- Face-to-face group (Active Comparator): This group underwent conventional face-to-face exercise.
  Interventions: Other: Face-to-face exercise

INTERVENTIONS:
Other: Tele-rehabilitation exercise — For this group, McKenzie extension exercises were applied to 50 patients online via the zoom platform.
  Arms: Tele-rehabilitation group
Other: Face-to-face exercise — For this group, 50 patients face-to-face in the clinical environment under the supervision of a physiotherapist in charge.
  Arms: Face-to-face group

SUMMARY:
The aim of this study was to investigate the effect of telerehabilitation on pain, disability, kinesiophobia and normal range of motion in patients with chronic non-specific low back pain. The study included 100 patients aged 18-64 years with chronic non-specific low back pain. In our study, McKenzie extension exercises were applied to 50 patients online via the zoom platform and to 50 patients face-to-face in the clinical environment under the supervision of a physiotherapist in charge. In our study, pain was assessed with the VAS, disability was assessed with the ODI, kinesiophobia was assessed with the TKS, and ROM was assessed with a goniometer. As a result of our study, there was no statistically significant difference in VAS values between both groups, a statistically significant difference was observed in both groups according to the measurement times and the pain level decreased in both groups. As a result of our study, there was no statistically significant difference in ODI values between both groups, a statistically significant difference was observed in both groups according to the measurement times and the level of disability decreased in both groups. As a result of our study, there was no statistically significant difference between the two groups in TKS values and no difference was observed according to the measurement times in both groups. As a result of our study, there was no statistically significant difference in ROM values between both groups, a statistically significant difference was observed in both groups according to the measurement times and ROM values increased. In conclusion, telerehabilitation in patients with chronic non-specific low back pain is as effective as face-to-face exercise training in improving pain, disability and range of motion levels, but the effect of telerehabilitation on improving kinesiophobia has not been found.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effect of telerehabilitation on pain, disability, kinesiophobia and normal range of motion in patients with chronic non-specific low back pain. The study included 100 patients aged 18-64 years with chronic non-specific low back pain. In our study, McKenzie extension exercises were applied to 50 patients online via the zoom platform and to 50 patients face-to-face in the clinical environment under the supervision of a physiotherapist in charge. In our study, pain was assessed with the Visual Analogue Scale (VAS), disability was assessed with the Oswestry Disability Index (ODI), kinesiophobia was assessed with the Tampa Kinesiophobia Scale (TKS), and Range of Motion (ROM) was assessed with a goniometer. As a result of our study, there was no statistically significant difference in VAS values between both groups (p>0.05), a statistically significant difference was observed in both groups according to the measurement times and the pain level decreased in both groups (p<0.05). As a result of our study, there was no statistically significant difference in ODI values between both groups (p>0,05), a statistically significant difference was observed in both groups according to the measurement times and the level of disability decreased in both groups (p<0,05). As a result of our study, there was no statistically significant difference between the two groups in TKS values (p>0,05) and no difference was observed according to the measurement times in both groups (p>0,05). As a result of our study, there was no statistically significant difference in ROM values between both groups (p>0.05), a statistically significant difference was observed in both groups according to the measurement times and ROM values increased (p<0.05). In conclusion, telerehabilitation in patients with chronic non-specific low back pain is as effective as face-to-face exercise training in improving pain, disability and range of motion levels, but the effect of telerehabilitation on improving kinesiophobia has not been found.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-64 years of age,
* Having non-specific low back pain for ≥3 months,
* Not having radicular symptoms related to low back pain

Exclusion Criteria:

* History of surgery on the spine and/or extremities,
* Diagnosis of malignancy,
* Orthopaedic and neurological disorders affecting the evaluation and treatment, - Psychiatric illness,
* Physical therapy for low back pain in the last six months,
* Being pregnant.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Disability | 18 months
  In our study, disability has assessed with the Oswestry Disability Index (ODI).
Pain intensity | 18 months
  In our study, pain has assessed with the Visual Analogue Scale (VAS). Scores range from 0 to 10
Kinesiophobia | 18 months
  In our study, kinesiophobia has assessed with the Tampa Kinesiophobia Scale (TKS). Scores range from 17 to 68 points.

SECONDARY OUTCOMES:
Range of motion | 18 months
  In our study, Range of Motion (ROM) has assessed with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Demirguc, PhD, Professor, Study Director — Sanko University
Locations (1):
- Sanko University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The publication of the scientific article in a journal might be shared with other researchers.